CLINICAL TRIAL: NCT04197271
Title: Management of Acutely Symptomatic Hernia: An Observational Study
Brief Title: Management of Acutely Symptomatic Hernia
Acronym: MASH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20908
Record Dates: First submitted 2019-09-09; First posted 2019-12-13 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hernia; Emergencies; Surgery--Complications
Keywords: outcome; hernia; emergency
MeSH Terms: conditions — Hernia; Emergencies | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acutely symptomatic abdominal wall hernia: Patients presenting to emergency surgical services with acutely symptomatic abdominal wall hernia (excluding parastomal).
  Interventions: Procedure: Emergency Hernia Repair; Other: Conservative management

INTERVENTIONS:
Procedure: Emergency Hernia Repair — Emergency repair of hernia using method selected by treating surgeon.
Other: Conservative management — Treatment of hernia without resort to surgery
  Other Names: Non-operative management

SUMMARY:
Acutely symptomatic abdominal wall hernia can cause many symptoms and complications. They can be associated with levels of morbidity beyond that seen in emergency laparotomy. There is limited data to guide practice in this field. This observational cohort study will explore variation in practice around assessment, repair and outcomes of hernias treated in the emergency setting.

DETAILED DESCRIPTION:
There are many different types of hernia, with the most common being in the groin or at the umbilicus. Hernias affect a significant proportion of the population and can vary from producing no symptoms at all, to causing a blockage to the bowel that requires urgent surgery. Hernias affect people of all ages and degrees of health, but become increasingly common with age. As our population ages and therefore becomes generally more unwell, the risks of surgery increase. Recent evidence suggests that emergency hernia repair is associated with worse outcomes than planned procedures. At present there are limited guidelines for the management of acutely symptomatic hernias and therefore practice varies between hospitals.

This cohort study will capture information on patients treated in the UK for acutely symptomatic hernia, and will provide information on variation in assessment, and technical aspects of repair. It will also capture health utility data out to 90 days post discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients admitted directly to the emergency surgery service (via A+E or GP)
* Patients referred to the emergency surgical team by another inpatient specialty
* Patients with a diagnosis of an acutely symptomatic hernia made by a specialist surgical trainee (ST3+) or Consultant Surgeon
* Willing to take part in the study

Exclusion Criteria:

* Patients under 18 years of age
* Pregnant women
* Patients with a symptomatic parastomal, hiatal or diaphragmatic hernia
* Patients with a traumatic hernia
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified from attendance at UK hospitals which provide emergency surgical services.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-24 (Estimated)

PRIMARY OUTCOMES:
In hospital morbidity | up to 28 days after surgery
  As defined using the comprehensive complication index

SECONDARY OUTCOMES:
Mortality | Measured at baseline, 30 days post discharge, and 90 days post recruitment
  Death occuring (binary)
Hospital length of stay | Within 30 days of recruitment to study
  Time from admission to discharge measured in days
Unplanned readmission within 30 days | Up to 30 days of recruitment
  Unplanned readmission to hospital for any reason following treatment of hernia
Change in health utility | Measured at baseline, 30 days post discharge and 90-days post recruitment
  Measured using EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Lee, MRCS PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proctor VK, O'Connor OM, Burns FA, Green S, Sayers AE, Hawkins DJ, Smart NJ, Lee MJ; MASH Collaborators. Surgical site infections after emergency hernia repair: substudy from the Management of Acutely Symptomatic Hernia (MASH) study. BJS Open. 2023 Jan 6;7(1):zrac155. doi: 10.1093/bjsopen/zrac155. PMID 36633418